CLINICAL TRIAL: NCT04535518
Title: Efficacy of Primary Treatment With Immunoglobulin Plus Infliximab for the Early Regression of Coronary Artery Lesion in Kawasaki Disease: a Multicenter, Open-label, Blinded-end Randomized Controlled Study.
Brief Title: Efficacy of Immunoglobulin Plus Infliximab for the Early Regression of Coronary Artery Lesion in Kawasaki Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Children's Hospital (Other); Shanghai Children's Medical Center (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai 10th People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KD-4-01
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Kawasaki Disease
Keywords: Kawasaki disease; infliximab; coronary artery lesion
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Immunoglobulins, Intravenous; Aspirin; Infliximab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants and physicians will not be masked to the assignment. Pediatric cardiologists who assess coronary artery lesions (CAL) by echocardiography will be masked to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the standard group (Active Comparator): 1. IVIG 2 g/kg once, given within 12 to 24 hours;
  2. Aspirin 30 mg/kg in oral per day (given in 3 divided doses), then 3 to 5 mg/kg per day when fever subsides for 72 hours and C-reactive protein (CRP) is normal. Aspirin will be continued for at least 6 weeks after onset of illness.
  Interventions: Drug: IVIG; Drug: Aspirin
- the standard + infliximab group (Experimental): 1. IVIG 2 g/kg once, given within 12 to 24 hours;
  2. Aspirin 30 mg/kg in oral per day (given in 3 divided doses), then 3 to 5 mg/kg per day when fever subsides for 72 hours and C-reactive protein (CRP) is normal. Aspirin will be continued for at least 6 weeks after onset of illness.
  3. Intravenous infliximab at single dose of 5 mg/kg, given more than 2 hours.
  Interventions: Drug: IVIG; Drug: Aspirin; Drug: Infliximab

INTERVENTIONS:
Drug: IVIG — IVIG at a single dose of 2 g/kg
  Other Names: Intravenous Immunoglobulins, Human
Drug: Aspirin — Aspirin 30 mg/kg in oral per day (given in 3 divided doses), then 3 to 5 mg/kg per day when fever subsides for 72 hours and C-reactive protein (CRP) is normal. Aspirin will be continued for at least 6 weeks after onset of illness.
  Other Names: Acetylsalicylic acid
Drug: Infliximab — Intravenous infliximab at single dose of 5 mg/kg, given more than 2 hours.
  Other Names: Remicade
  Arms: the standard + infliximab group

SUMMARY:
This study evaluates the efficacy of the addition of infliximab to conventional initial treatment (intravenous immunoglobulin [IVIG] plus aspirin) in early regression of coronary artery lesion in patients with Kawasaki disease (KD).

DETAILED DESCRIPTION:
This is a multicenter, open-label, blind-end, randomized controlled trial at 5 hospitals in Shanghai, China. The KD children diagnosed within 14 days of onset according to the diagnostic criteria for KD released by American Heart Association (AHA) in 2017 will be considered for participants in the trial. The patients meeting eligibility criteria will be randomly assigned in a 1:1 ratio to the control group (receiving 2 g/kg*1 IVIG and 30 mg/kg/d aspirin) or intervention group (receiving 2 g/kg*1 IVIG, 30 mg/kg/d aspirin and additional 5 mg/kg*1 infliximab) based on the randomly block design (block sizes 4). Baseline characteristics of each participant will be collected, including sex, age of onset, height, body weight, subtype of KD, fever days before initial IVIG, other clinical manifestations, echocardiographic findings at enrolment, and a series of pre-IVIG laboratory tests. Two-dimensional echocardiography will be performed at least 7 timepoints: at admission, 2 weeks, 1 month, 3 months, 6 months, 9 months and 12 months after onset of KD to assess the coronary artery lesions.

ELIGIBILITY:
Inclusion Criteria:

* Meeting diagnostic criteria for KD released by American Heart Association (AHA) in 2017, including complete KD (also sometimes referred to as typical or classic KD) and incomplete KD ((also sometimes referred to as atypical KD);
* Diagnosed within 14 days of illness (including the 14th day, considering the first day of illness as the first day of fever);
* Not treated with IVIG or other treatments for KD yet;
* Z score of any coronary artery of LMCA, LAD, LCX, the proximal and middle segment of RCA ≥ 2 calculated based on the height, weight and coronary artery diameter measured by echocardiography;
* Aged between one month and 14 years.

Exclusion Criteria:

* Receiving steroids or other immunosuppressive agents in the previous 30 days;
* With a previous history of KD;
* Afebrile and all the inflammation indicators (including white blood cell count, CRP, and erythrocyte sedimentation) become normal before enrolment;
* With suspected infectious diseases including tuberculosis, sepsis, septic meningitis, peritonitis, bacterial pneumonia, varicella, influenza, EBV infection, etc;
* With serious immune diseases such as immunodeficiency or chromosomal abnormalities;
* Unable to be followed up for at least 1 year.

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of the regression of coronary artery lesion (CAL) at one month of illness | at one month of illness
  The regression of CAL is defined as z < 2 of all coronary arteries of LMCA, LAD, LCX, and the proximal and middle segment of the RCA.Two-dimensional echocardiography will be performed to evaluate CAL at 1 month of illness. The measurement of each patient included the diameter of the left main coronary artery (LMCA), the left anterior descending artery (LAD), the left circumflex coronary artery (LCX), and the proximal and middle segments of the right coronary artery (RCA). Z score of each coronary artery will be calculated (Journal of the American Society of Echocardiography, 2011, 24(1):60-74).

SECONDARY OUTCOMES:
Percentage of the need for additional treatment | from admission to discharge (about 2 weeks of illness)
  Participants who have recurrent or persistent fever (axillary temperature ≥37.5°C or rectal temperature ≥38°C) after 36 hours of completion of initial IVIG infusion will be given additional treatment, including a second dose of IVIG (2 g/kg), or a high dose of methylprednisolone (10 to 30 mg/kg per day), or other immunosuppressive agents such as ciclosporin and cyclophosphamide, or a combination with two or more drugs, or even more aggressive treatment such as plasmapheresis, depending on patients'condition and physicians' experience. Axillary temperature (or rectal temperature) will be measured every 6 hours a day during hospitalization.
z scores of LMCA throughout the study period | from admission to 12 months of illness
  This is a repeated measurement. Z score will be calculated based on the height, weight and coronary artery diameter (Journal of the American Society of Echocardiography, 2011, 24(1): 60-74.). The internal diameter of LMCA will be measured by echocardiography at least seven time points: at enrollment, at 2 weeks, 1 month, 3 months, 6 months, 9 months and 12 months of illness.
z scores of LAD throughout the study period | from admission to 12 months of illness
  This is a repeated measurement. Z score will be calculated based on the height, weight and coronary artery diameter (Journal of the American Society of Echocardiography, 2011, 24(1): 60-74.). The internal diameter of LAD will be measured by echocardiography at least seven time points: at enrollment, at 2 weeks, 1 month, 3 months, 6 months, 9 months and 12 months of illness.
z scores of LCX throughout the study period | from admission to 12 months of illness
  This is a repeated measurement. Z score will be calculated based on the height, weight and coronary artery diameter (Journal of the American Society of Echocardiography, 2011, 24(1): 60-74.). The internal diameter of LCX will be measured by echocardiography at least seven time points: at enrollment, at 2 weeks, 1 month, 3 months, 6 months, 9 months and 12 months of illness.
z scores of the proximal segment of RCA throughout the study period | from admission to 12 months of illness
  This is a repeated measurement. Z score will be calculated based on the height, weight and coronary artery diameter (Journal of the American Society of Echocardiography, 2011, 24(1): 60-74.). The internal diameter of the proximal segment of RCA will be measured by echocardiography at least seven time points: at enrollment, at 2 weeks, 1 month, 3 months, 6 months, 9 months and 12 months of illness.
z scores of the middle segment of RCA throughout the study period | from admission to 12 months of illness
  This is a repeated measurement. Z score will be calculated based on the height, weight and coronary artery diameter (Journal of the American Society of Echocardiography, 2011, 24(1): 60-74.). The internal diameter of the middle segment of RCA will be measured by echocardiography at least seven time points: at enrollment, at 2 weeks, 1 month, 3 months, 6 months, 9 months and 12 months of illness.
Duration of fever (hours) after initiation of initial IVIG infusion | from initiation of initial IVIG infusion to the first record of being afebrile (defined as an axillary temperature <37.5 for more than 24 hours)
  Participants with an axillary temperature <37.5℃ (or rectal temperature <38℃) for more than 24 hours are considered afebrile. Axillary temperature (or rectal temperature) will be measured every 6 hours a day during hospitalization. Record the time of the initiation of IVIG infusion and the time of the body temperature first becoming normal.
Change in serum C-reactive protein (CRP) concentration | from admission to 72 hours after completion of initial IVIG infusion
  CRP level is measured before initial IVIG infusion and 72 hours after completion of initial IVIG infusion.Change would be described by difference.
Number of patients with serious adverse events | from admission to 12 months of illness
  This is a composite outcome, including death, hypertension (defined as the blood pressure (BP) ≥90th percentile for age and height or ≥ 120/80 mmHg in the children younger than 13, and ≥ 120/80 mmHg in children ≥ 13 years), severe infection (such as septicopyemia, pulmonary infection and urinary system infection), allergic reactions, heart failure, thrombosis, etc.
Percentage of the regression of coronary artery lesion (CAL) at 3 months of illness | at 3 months of illness
  The regression of CAL is defined as the z < 2 of all coronary arteries of LMCA, LAD, LCX, and the proximal and middle segment of the RCA.
Percentage of the regression of coronary artery lesion (CAL) at 6 months of illness | at 6 months of illness
  The regression of CAL is defined as the z < 2 of all coronary arteries of LMCA, LAD, LCX, and the proximal and middle segment of the RCA.
Percentage of the regression of coronary artery lesion (CAL) at 9 months of illness | at 9 months of illness
  The regression of CAL is defined as the z < 2 of all coronary arteries of LMCA, LAD, LCX, and the proximal and middle segment of the RCA.
Percentage of the regression of coronary artery lesion (CAL) at 12 months of illness | at 12 months of illness
  The regression of CAL is defined as the z < 2 of all coronary arteries of LMCA, LAD, LCX, and the proximal and middle segment of the RCA.

CONTACTS AND LOCATIONS:
Overall Officials: Guoying Huang, MD., Study Director — Children's Hospital of Fudan University
Locations (5):
- China (5):
  - Shanghai Children's Hospital, Shanghai
  - Shanghai 10th People's Hospital, Shanghai
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Children's Medical Center, Shanghai
  - Children's Hospital of Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dallaire F, Dahdah N. New equations and a critical appraisal of coronary artery Z scores in healthy children. J Am Soc Echocardiogr. 2011 Jan;24(1):60-74. doi: 10.1016/j.echo.2010.10.004. Epub 2010 Nov 13. PMID 21074965